CLINICAL TRIAL: NCT06557980
Title: Effectiveness of Calcium Silicate and Sodium Fluoride Nanoparticles in The Management of Dentin Hypersensitivity (Randomized Controlled Clinical Trial and In-Vitro Study)
Brief Title: Effectiveness of Calcium Silicate and Sodium Fluoride Nanoparticles in The Management of Dentin Hypersensitivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Kareem Abd El Hamid Lotfy, Assistant Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hypersensitivity management
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Toothpastes

STUDY DESIGN:
Intervention Model Description: Each toothpaste will be applied uniformly twice per day (morning and bed time) to the hypersensitive surfaces for30 seconds. After that, the patient will rinse their mouth with plain water.
  Responses to the various stimuli will be evaluated using the same tactile and thermal stimuli used previously, and scores will be recorded 1day1,2 ,4 ,8 ,12 , weeks then 6 and 12 months after their application, respectively.
  Furthermore, the patients will be advised to report to the operator any unanticipated pain seizures, erroneous usage as well as the number of applications of a specific desensitizing agent required to elicit a positive response will also be recorded. The results will be statistically analyzed after 8 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The operator, the assessor as well as the data analyst will be blinded to material assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toothpaste containing calcium silicate nanoparticles (Active Comparator): patients with hypersensitive areas will use the calcium silicate based toothpaste
  Interventions: Other: toothpaste
- Toothpaste containing sodium fluoride nanoparticles (Active Comparator): patients with hypersensitive areas will use the sodium fluoride based toothpaste
  Interventions: Other: toothpaste

INTERVENTIONS:
Other: toothpaste — group of patients with hypersensitive areas will use the calcium silicate toothpaste twice per day (morning and bedtime) the toothpaste will be applied uniformly using medium toothbrush to the hypersensitive surfaces for 30seconds. After that, the patient will rinse their mouth with plain water. the other group of patients will use the sodium fluoride toothpaste twice per day (morning and bedtime). The toothpaste will be applied uniformly using a medium toothbrush to the hypersensitive areas for 30 seconds after that the patients will rinse their mouth with plain water

SUMMARY:
This study will be performed to assess the effect of inert prepared tooth paste loaded with Calcium Silicate Nanoparticles (CSNPs) and compare it to another one containing Sodium Fluoride Nanoparticles in the management of patients complaining of hypersensitivity and laboratory investigating the efficacy of CSNPs and NaFl Nps containing toothpaste in dentinal tubules occlusion.

DETAILED DESCRIPTION:
Hypersensitivity has been defined as the pain arising from exposed dentin, typically in response to chemical, thermal, tactile or osmotic stimuli that cannot be explained as arising from any other form of dental defect or pathology. The pain of dentin hypersensitivity is classically, short, sharp, of rapid onset in character and of the duration of the applied stimuli. hypersensitivity was first documented by Blum. Although much has been learnt about hypersensitivity overtime, yet the mechanism of pain was explained by several hypotheses welling to be aware about the nature of the Disease firstly was the hypothesis that dentin was innervated and therefore, nerves were directly triggered by the stimulus. A further theory, termed the odontoblast transducer mechanism. Currently, the most widely accepted theory is the hydrodynamic theory which determined that there was an outward flow of fluid along the dentinal tubules.

In addition to extrapolation of the pain mechanism, allocating the etiology and the risk factors have a crucial impact on the disease outcome as well as the line of treatment. For hypersensitivity to occur lesion localization, where the dentin surface of a tooth must be exposed. And a lesion initiation must take place where the number of dentin tubules in close proximity to each other must be patent from the pulp to the oral environment.

Several in vitro and in situ data, case report data and epidemiological surveys summarized the most common etiologic and risk factors in the two main causes: gingival recession exposing dentin, either by periodontal Disease, zealous brushing, smoking and loss of hard tissue exposing dentin, also by frank carious lesions with dentin exposure of smooth tooth surface or development of non-carious cervical lesions.

Eventually based on the great knowledge about hypersensitivity nature, Etiologic and risk factors the dental professionals can now select the appropriate line of treatment either with conservative non-surgical intervention ex; Elimination of etiological factors, addition of desensitizers to toothpastes like Potassium nitrate, Strontium, Arginine and Calcium Carbonate, Calcium Sodium Phosphosilicate. Use of Dentin desensitizing products which have different ingredients, such as fluoride, hydroxyethyl methacrylate, glutaraldehyde, oxalate and potassium nitrate, as well as a combination of these ingredients.

Several in vitro, in situ as well as in vivo studies tackled the immense remineralizing capabilities of calcium silicate and it's in vitro promising results in formation of hydroxyapatite on enamel as well as occluding dentinal tubules thus giving potential anti-hypersensitivity benefits. However in vivo anti-hypersensitivity benefits were not tackled enough in literature.

This study will be performed to clinically assess the effect of toothpaste loaded with calcium silicate Nanoparticles (CS NPs) and compare it to one loaded with Sodium fluoride Nanoparticles (NaFL NPs) in the management of dentin hypersensitivity and laboratory investigating their efficacy in dentinal tubules occlusion. The null Hypothesis is the CS NPs has the same effect as Na FLNPs in the management of hypersensitivity complaining patient. The alternative hypothesis is the dentinal tubules occlusion by CSNPs will be like that one produced by Na FLNPs.

ELIGIBILITY:
Inclusion Criteria:

* Hypersensitive areas on facial surfaces of the teeth (incisors, cuspids, bicuspids, and first molars with exposed cervical dentine)
* Areas with hard tissue erosion
* cuneiform defect, pathological abrasion.
* Gingival recession
* Good overall physical health
* Age between 20 to 40 years; and provision of written informed consent

Exclusion Criteria:

* chipped teeth
* Defective restorations
* fractured un displaced cuspids
* deep dental caries
* deep periodontal pockets
* orthodontic appliances, dentures, or bridgework that would interfere with the evaluation of hypersensitivity.
* periodontal surgery within the previous 6 months.
* ongoing treatment with antibiotics and/or anti-inflammatory and/or analgesic drugs.
* ongoing treatment for tooth hypersensitivity, pregnancy, or lactation; heavy smoking and alcohol or drug abuse.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The Visual analogue scale | one year
  The Visual analogue scale on a scale (0 = no pain,10 = extreme pain).
The Verbal rating scale | one year
  The Verbal rating scale from to: (0 = no discomfort, 1=mild discomfort,2 = significant discomfort,3= significant discomfort lasting more than 10 seconds)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: for anyone